CLINICAL TRIAL: NCT05629104
Title: Biological Valve Prosthesis in Aortic Stenosis - Imaging, Biomarkers, Physical Performance and Patient Related Factors Predictive to Long-term Outcome (Bio-AS)
Brief Title: Prediction of Long-term Outcome in Aortic Stenosis After Valve Intervention
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: Bio-AS
Record Dates: First submitted 2020-07-17; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preserved heart function: The group will be defined as preserved left ventricular ejection fraction (LVEF) with and without hypertrophy and with and without reduced global longitudinal strain (GLS).
  Interventions: Other: There is no intervention since it is an observational study patients are treated according to clinical praxis
- Reduced heart function: The group will be defined as reduced LVEF
  Interventions: Other: There is no intervention since it is an observational study patients are treated according to clinical praxis

INTERVENTIONS:
Other: There is no intervention since it is an observational study patients are treated according to clinical praxis — No intervention

SUMMARY:
Patients with severe aortic stenosis accepted for transcatheter intervention or open surgery are included before the intervention, and then followed up with clinical visits during the first year after intervention. Imaging with echocardiography and computed tomography (CT) are performed together with additional imaging with magnetic resonance imaging (MRI) and Positron emissions tomography (PET)-CT in a subgroup of the study population. Blood samples, physical performance and questionnaires with focus on frailty and heart failure are also collected at each visit. A follow up with information of the outcomes after 2-5 years will be performed through national registries.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for aortic valve intervention

Exclusion Criteria:

* No able to follow the study protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients accepted for aortic valve intervention due to aortic stenosis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Semiquantitative assessment of protein levels associated with myocardial performance | One year after intervention.
  Level of normalized protein expression (NPX) in plasma, assessed by a multiplex proximity extension assay panel (Olink Bioscience, Uppsala, Sweden).
Imaging parameters associated with clinical outcome after intervention | One year after intervention
  Global longitudinal strain (%) of the right and left ventricle. The clinical outcome defined as a combination of mortality and hospitalization of heart failure
Semiquantitative assessment of protein levels associated with myocardial performance associated with clinical outcome after intervention | Two years after intervention
  Level of normalized protein expression (NPX) in plasma, assessed by a multiplex proximity extension assay panel (Olink Bioscience, Uppsala, Sweden). The clinical outcome defined as a combination of mortality and hospitalization for heart failure.

SECONDARY OUTCOMES:
Imaging parameters associated with clinical outcome after intervention | Two years after intervention
  Volumes of the right and left ventricle (mL/m2). The clinical outcome defined as a combination of mortality and hospitalization for heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Christersson, MD PhD, Principal Investigator — VO hjärt-lungmedicin och klinisk fysiologi Akademiska Sjukhuset
Locations (1):
- Department of cardiology Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No